CLINICAL TRIAL: NCT00589810
Title: Whole Genome Association Study to Identify and Validate Genes for Restenosis: CardioGene Validation Proposal
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Stephen G. Ellis, M.D., Principal Investigator, The Cleveland Clinic
Other Study IDs: 06-887
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Coronary Restenosis
Keywords: ISR; in-stent restenosis; restenosis; BMS; bare metal stent; revascularization; genetic; cardiac catheterization
MeSH Terms: conditions — Coronary Restenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Controls: Controls = Patients in Genebank that had BMS placed that did not go on to have ISR within 1 year of BMS placement and have not had prior ISR in any vessel ever. If testing is available, the Control status will be further verified by angiographic documentation of <50% luminal loss with the stent or negative stress test six or more months after stenting.
- Cases: Cases = Patients in Genebank that had BMS placed that went on to have ISR which is defined as PCI or CABG to the Target Vessel within 1 year of the BMS placement.

SUMMARY:
In this replication study at the Cleveland Clinic, we seek to collaborate to validate findings of the CardioGene Study in an independent cohort of patients who have undergone bare metallic stenting.

DETAILED DESCRIPTION:
Dr. Elizabeth Nabel, Dr. Santhi K. Ganesh and colleagues at the National Institutes of Health have completed a genetic association study, entitled the CardioGene Study, using 100,000 SNPs spanning the entire human genome in subjects with restenosis after percutaneous intervention using bare metallic stents (Ganesh SK, 2004). In this replication study at the Cleveland Clinic, we seek to collaborate to validate findings of the CardioGene Study in an independent cohort of patients who have undergone bare metallic stenting. This study will examine samples and clinical data collected of subjects undergoing cardiac catheterization who meet study criteria, selected from the GeneBank. In the Genebank repository, subjects are informed their samples may be used indefinitely for study and consent to having their data/samples shared with other investigators at the Cleveland Clinic or other collaborating institutions. No information that might identify subjects is shared with collaborating investigators and samples will be shared in a de-identified manner, using assigned study numbers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 with informed consent for participation in Genetics Research
* BMS placed in a de novo(previously untreated by any type of PCI) lesion within a native coronary artery (not within a bypass graft) lesion
* Outcome data available at 12 months

Exclusion Criteria:

For both cases and controls:

* Age less than 18
* No informed consent for Genetic Research
* BMS placed in a bypass graft.
* Radiation to the same lesion treated with bare metal stent at the time of index stenting (continued on next page)
* A drug-eluting stent within or overlapping the target lesion BMS placed at the time index stenting.
* Participation in a cardiovascular study at any time between index stenting procedure and day 365 post stenting or until TVR, which ever occurs first, which meets one or more of the following:

  * Placebo vs an active drug being studied against restenosis rates, atheroma volume or thrombosis, in which unblinding information is not available and the study results are unknown or the active drug is shown to have a positive effect.
  * Placebo vs active drug known to have an effect on restenosis rates, atheroma volume or thrombosis in which unblinding information is not available.
  * Blinded randomized studies involving two classes of drug in which the results are unknown or the results of the study show superiority to one of the treatment arms and unblinding information is not available.

For controls only: in addition to the exclusions above:

* any prior history of TVR(TRRS)
* positive stress test or cath with > or equal to 50% stenosis of target lesion within one year of index bare metal stenting.
* Subjects reported to be deceased in the Interventional Registry or through chart abstraction without negative cath results or negative stress test results between 5 months and 13 months post index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cleveland Clinic patients already enrolled in the GeneBank study who have had left heart catheterization and bare metal stenting
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
In-stent restenosis | 1 year

SECONDARY OUTCOMES:
Target vessel revascularization | 1 year
Positive stress test | 1 year
Negative cardiac catheterization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ellis, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stone GW, Ellis SG, Cox DA, Hermiller J, O'Shaughnessy C, Mann JT, Turco M, Caputo R, Bergin P, Greenberg J, Popma JJ, Russell ME; TAXUS-IV Investigators. A polymer-based, paclitaxel-eluting stent in patients with coronary artery disease. N Engl J Med. 2004 Jan 15;350(3):221-31. doi: 10.1056/NEJMoa032441. PMID 14724301
- [Background] Sousa JE, Costa MA, Abizaid AC, Rensing BJ, Abizaid AS, Tanajura LF, Kozuma K, Van Langenhove G, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Sustained suppression of neointimal proliferation by sirolimus-eluting stents: one-year angiographic and intravascular ultrasound follow-up. Circulation. 2001 Oct 23;104(17):2007-11. doi: 10.1161/hc4201.098056. PMID 11673337
- [Background] Sousa JE, Costa MA, Abizaid A, Abizaid AS, Feres F, Pinto IM, Seixas AC, Staico R, Mattos LA, Sousa AG, Falotico R, Jaeger J, Popma JJ, Serruys PW. Lack of neointimal proliferation after implantation of sirolimus-coated stents in human coronary arteries: a quantitative coronary angiography and three-dimensional intravascular ultrasound study. Circulation. 2001 Jan 16;103(2):192-5. doi: 10.1161/01.cir.103.2.192. PMID 11208675
- [Background] Schaid DJ. Power and sample size for testing associations of haplotypes with complex traits. Ann Hum Genet. 2006 Jan;70(Pt 1):116-30. doi: 10.1111/j.1529-8817.2005.00215.x. PMID 16441261
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Lowe HC, Oesterle SN, Khachigian LM. Coronary in-stent restenosis: current status and future strategies. J Am Coll Cardiol. 2002 Jan 16;39(2):183-93. doi: 10.1016/s0735-1097(01)01742-9. PMID 11788206
- [Background] Kastrati A, Schomig A, Elezi S, Schuhlen H, Dirschinger J, Hadamitzky M, Wehinger A, Hausleiter J, Walter H, Neumann FJ. Predictive factors of restenosis after coronary stent placement. J Am Coll Cardiol. 1997 Nov 15;30(6):1428-36. doi: 10.1016/s0735-1097(97)00334-3. PMID 9362398
- [Background] Ganesh SK, Skelding KA, Mehta L, O'Neill K, Joo J, Zheng G, Goldstein J, Simari R, Billings E, Geller NL, Holmes D, O'Neill WW, Nabel EG. Rationale and study design of the CardioGene Study: genomics of in-stent restenosis. Pharmacogenomics. 2004 Oct;5(7):952-1004. doi: 10.1517/14622416.5.7.949. PMID 15469413